CLINICAL TRIAL: NCT03558139
Title: A Phase 1b Trial of Hu5F9-G4 in Combination With Avelumab in Solid Tumor Patients and Checkpoint-Inhibitor-Naive Ovarian Cancer Patients Who Progress Within 6 Months of Prior Platinum Chemotherapy
Brief Title: Study of Magrolimab (Hu5F9-G4) in Combination With Avelumab in Solid Tumor Participants and Checkpoint-Inhibitor-Naive Ovarian Cancer Participants Who Progress Within 6 Months of Prior Platinum Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5F9006
Record Dates: First submitted 2018-05-30; First posted 2018-06-15 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — magrolimab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) (Experimental): Participants with solid tumors will be treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 30 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 15, 22, and 29 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 will consist of 35 days and Cycle 2 and subsequent cycle will consist of 28 days. Avelumab will be administered 1 hour prior to magrolimab infusion on days when both are given. Treatment will be administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
  Interventions: Drug: Magrolimab; Drug: Avelumab
- Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) (Experimental): Participants with solid tumors will be treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 will consist of 35 days and Cycle 2 and subsequent cycle will consist of 28 days. Avelumab will be administered 1 hour prior to magrolimab infusion on days when both are given. Treatment will be administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
  Interventions: Drug: Magrolimab; Drug: Avelumab
- Magrolimab 45 mg/kg + Avelumab 800 mg (Part 2, Ovarian Cancer Expansion) (Experimental): Participants with checkpoint inhibitor-naïve ovarian cancer will be treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 will consist of 35 days and Cycle 2 and subsequent cycle will consist of 28 days. Avelumab will be administered 1 hour prior to magrolimab infusion on days when both are given. Treatment will be administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
  Interventions: Drug: Magrolimab; Drug: Avelumab

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: Hu5F9-G4
Drug: Avelumab — Administered intravenously
  Other Names: BAVENCIO®

SUMMARY:
The primary objectives of this study are to investigate the safety and tolerability of magrolimab in combination with avelumab in participants with advanced solid tumors and to confirm the safety and tolerability of this combination and evaluate the anti-tumor activity in participants with checkpoint inhibitor-naive ovarian cancer, fallopian tube cancer, and primary peritoneal carcinoma who have previously progressed within 1-6 months of receiving platinum chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Safety Run-in Cohort: Pathologically confirmed advanced solid tumors.
* Ovarian Cancer Expansion Cohort: Histologically or cytologically confirmed, epithelial ovarian, fallopian tube, or peritoneal cancer.

  * Checkpoint inhibitor naive participants.
  * Willing to consent to 1 mandatory pre-treatment and 1 on-treatment tumor biopsy.
* Adequate performance status. Adequate hematological, liver, and kidney functions.
* Availability of pre-treatment tumor tissue to evaluate programmed cell death-ligand 1(PD-L1) expression.

Key Exclusion Criteria:

* Individuals with symptomatic or untreated central nervous system (CNS) metastases.
* Prior treatment with cluster of differentiation 47 (CD47) or signal regulatory protein alpha (SIRPα) targeting agents.
* Known active or chronic hepatitis B or C infection or human immunodeficiency virus (HIV).
* Red blood cell transfusion dependence.
* Prior organ transplantation requiring immunosuppression or active autoimmune disease.
* Significant medical diseases and/or history of uncontrolled intercurrent illness or other serious medical condition.
* Pregnancy or active breast feeding.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - University of Chicago, Chicago, Illinois
  - START Midwest, Grand Rapids, Michigan
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lakhani NJ, Patnaik A, Liao JB, et al. A phase 1b study of the anti-CD47 antibody magrolimab with the PD-L1 inhibitor avelumab in solid tumor & ovarian cancer patients [Abstract]. American Society of Clinical Oncology (ASCO)-Society for Immunotherapy of Cancer (SITC) Clinical Immuno-Oncology Symposium; 2020 06-08 February. Orlando, FL.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT03558139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 23 May 2018. The last study visit occurred on 03 December 2020.
Pre-assignment Details: 43 participants were screened.
Groups:
- Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in): Participants with solid tumors were treated with starting priming dose of 1 mg/kg of body weight magrolimab intravenous (IV) infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 30 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 15, 22, and 29 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days. Avelumab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
- Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in): Participants with solid tumors were treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1 and Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days. Avelumab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
- Magrolimab 45 mg/kg + Avelumab 800 mg (Part 2, Ovarian Cancer Expansion): Participants with checkpoint inhibitor-naïve ovarian cancer were treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days. Avelumab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
Period: Overall Study
Arm/Group | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 2, Ovarian Cancer Expansion)
Started | 6 | 7 | 21
Completed (One participant withdrew the consent and died after the last dose of study drug. The primary reason for study discontinuation was considered as "Consent Withdrawn".) | 0 | 0 | 0
Not Completed | 6 | 7 | 21
Not completed — Consent Withdrawn | 1 | 1 | 4
Not completed — Death | 5 | 3 | 8
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Study Ended Per Protocol | 0 | 3 | 6

BASELINE CHARACTERISTICS:
Population: All Treated participants included all participants who received at least 1 dose of any study drugs.
Groups:
- Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in): Participants with solid tumors were treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 30 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 15, 22, and 29 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days. Avelumab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
- Total: Total of all reporting groups
Arm/Group | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 2, Ovarian Cancer Expansion) | Total
Number analyzed (Participants) | 6 | 7 | 21 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (14.34) | 65.3 (7.48) | 64.5 (5.59) | 64.8 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 21 | 29
  Male | 2 | 3 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 5 | 7 | 18 | 30
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 7 | 20 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
CD68 Macrophages [Mean (Full Range); unit: cells] — Population: The data for mean baseline CD68 macrophage was not collected for participants in Part 1, Safety Run-in Cohorts. Data are reported for the participants who enrolled in Ovarian Cancer Expansion Cohort (Part 2) and for whom paired biopsies were available.
  cells
    number analyzed (Participants) | 0 | 0 | 6 | 6
    (all) |  |  | 6.3 [3.00 to 10.00] | 6.3 [3.00 to 10.00]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) in Safety Run-in (Part 1)
Description: A DLT was defined as a ≥ Grade 3 AE that was assessed as related to either magrolimab or avelumab that occurred during the 5-week DLT assessment period with protocol-defined allowed exceptions. Any treatment-emergent adverse event (TEAE) that was, in the opinion of the Clinical Trial Steering Committee, of potential clinical significance such that further dosing exposed participants to unacceptable risk, was considered a DLT.
Time Frame: From the first dose date up to 5 weeks
Population: DLT evaluable participants: Participants in the Safety Run-in Part who met if either of the following criteria during the DLT assessment period:
  * the participant experienced a DLT at any time after initiation of the first infusion of either magrolimab or avelumab and during the 5-week DLT assessment period
  * the participant completed at least 4 (or 5 if assigned to magrolimab 45 mg/kg + avelumab 800 mg) infusions of magrolimab at the assigned dose and 2 infusions of avelumab.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in)
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. Treatment-emergent AEs were defined as those AEs that worsened or occurred during or after a participant's first dose of any study treatment and those existing AEs that worsened during the study and within 30 days after the last administration of any study treatment or initiation of subsequent anticancer therapy, whichever occurred first.
Time Frame: First dose date up to last dose plus 30 days (maximum treatment duration 18.3 months)
Population: All Treated participants (included all participants who received at least 1 dose of any study drugs) were analyzed. Per planned analysis, AE data were summarized by the magrolimab maintenance dose level. One participant in Part 2 received maintenance dose of 20 mg/kg. Because of confidentiality reason, data for this participant was not provided separately and included in "Magrolimab Priming Dose or Magrolimab 20 mg/kg" arm.
Measure: Number; unit: percentage of participants
Groups:
- Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in + Part 2, Ovarian Cancer Expansion): Participants with solid tumors (Part 1) or checkpoint inhibitor-naive ovarian cancer (Part 2) were treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1 and Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles. Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days. Avelumab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
- Magrolimab Priming Dose or Magrolimab 20 mg/kg: Participants who received only priming dose of magrolimab (1 mg/kg) in Part 2 of the study.
  For 1 participant (Part 2) magrolimab infusion was not completed at the first maintenance dose because of adverse event and <60% of planned dose was administered. Subsequently the participant was treated at 20 mg/kg dose level.
Arm/Group | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in + Part 2, Ovarian Cancer Expansion) | Magrolimab Priming Dose or Magrolimab 20 mg/kg
Number analyzed (Participants) | 6 | 25 | 3
percentage of participants | 100 | 100 | 100

3. Primary Outcome: Percentage of Participants With Objective Response (ORR) Assessed by Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 in Participants With Ovarian Cancer
Description: Objective response was defined as the percentage of participants with objective response which consisted of complete response (CR)+ partial response (PR) determined by RECIST v 1.1. CR: Disappearance of all target and all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (< 10 mm short axis). Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From screening until 26.2 months (assessed on Day 1 of Cycle 3 then every 2 cycles from Cycle 5 onwards up to 26.2 months; 1 cycle: 28 days)
Population: Efficacy Analysis Set included checkpoint inhibitor-naive participants with ovarian cancer, who had previously progressed within 6 months of receiving platinum chemotherapy and received at least one dose of magrolimab during this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Magrolimab 45 mg/kg + Avelumab 800 mg (Ovarian Cancer Participants): Participants with checkpoint inhibitor-naive ovarian cancer who previously progressed within 6 months of receiving platinum chemotherapy were treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days. Avelumab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
Arm/Group | Magrolimab 45 mg/kg + Avelumab 800 mg (Ovarian Cancer Participants)
Number analyzed (Participants) | 21
percentage of participants | 0.0 [0.0 to 16.8]

4. Secondary Outcome: Recommended Phase 2 Dose and Schedule (RP2DS) of Magrolimab in Combination With Avelumab
Description: The RP2DS was the dose of magrolimab in combination with avelumab with DLT rate less than 33% in at least 6 evaluable participants in Part 1. A DLT was defined as a ≥ Grade 3 AE that was assessed as related to either magrolimab or avelumab that occurred during the 5-week DLT assessment period with protocol-defined allowed exceptions. Any TEAE that was, in the opinion of the Clinical Trial Steering Committee, of potential clinical significance such that further dosing exposed participants to unacceptable risk, was considered a DLT.
Time Frame: From the first dose date up to 5 weeks
Population: All Treated participants in Part 1 were analyzed.
Measure: Number; unit: mg/kg
Groups:
- Magrolimab - Part 1 All Participants: Participants with solid tumors were treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 30 or 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) every 2 weeks on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
  Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days. Avelumab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until confirmed tumor progression, unacceptable toxicity, clinically significant change in the participant's status that precluded further treatment, voluntary withdrawal, or physician decision.
Arm/Group | Magrolimab - Part 1 All Participants
Number analyzed (Participants) | 13
mg/kg | 45

5. Secondary Outcome: Serum Concentrations of Magrolimab - Safety Run-in (Part 1)
Description: Serum concentrations will be drawn at pre-study drug infusion (within 12 hours) on Day (D) 1 and 22 in Cycle (C) 1; Days 1 and 15 in Cycle 2; Day 1 in Cycles 3 and 4; every 3rd cycle on Day 1 until Cycle 13; 1 hour post-magrolimab infusion on Days 1 and 8 in Cycle 1; 24 hours post magrolimab infusion (Part 1 only) on Days 1 and 8 in Cycle 1; pre-study drug infusion on Day 1 in Cycles 5 and 11 (Part 1 Magrolimab 45 mg/kg only); End of Treatment (EOT) visit (up to Cycle 13); Safety Follow-up Visit (30 days after last dose of magrolimab, maximum treatment duration 18.3 months). Cycle 1 consisted of 35 days and Cycle 2 and subsequent cycle consisted of 28 days.
Time Frame: Predose: (C1D1, C1D22, C2D1,C2D15, C3D1, C4D1, C5D1 [only for 45 mg/kg Part 1], C7D1, C10D1, C11D1 [only for 45 mg/kg Part 1], C13D1, EOT, Safety Follow-up); 1 hour postdose: (C1D1, C1D8); 24 hours postdose: (C1D1, C1D8)
Population: Pharmacokinetic Analysis Set (included participants who received any amount of magrolimab with at least one detectable post-treatment serum concentration of magrolimab) with available data in Part 1 were analyzed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in)
Number analyzed (Participants) | 6 | 7
ug/mL
  Pre-dose on Day 1 Cycle 1 | 0.00 (0.000) | 0.00 (0.000)
  1 hour post-magrolimab dose on Day 1 Cycle 1 | 0.76 (0.544) | 0.62 (0.583)
  24 hours post-magrolimab dose on Day 1 Cycle 1 | 0.06 (0.139) | 0.04 (0.104)
  1 hour post-magrolimab dose on Day 8 Cycle 1 | 925.83 (171.835) | 981.43 (249.861)
  24 hours post-magrolimab dose on Day 8 Cycle 1: number analyzed (Participants) | 5 | 7
  24 hours post-magrolimab dose on Day 8 Cycle 1 | 487.80 (108.493) | 680.57 (128.439)
  Pre-dose on Day 22 Cycle 1 | 403.50 (65.145) | 769.57 (209.417)
  Pre-dose on Day 1 Cycle 2: number analyzed (Participants) | 5 | 7
  Pre-dose on Day 1 Cycle 2 | 840.00 (155.259) | 867.57 (232.251)
  Pre-dose on Day 15 Cycle 2: number analyzed (Participants) | 5 | 7
  Pre-dose on Day 15 Cycle 2 | 447.20 (72.116) | 915.57 (295.178)
  Pre-dose on Day 1 Cycle 3: number analyzed (Participants) | 5 | 4
  Pre-dose on Day 1 Cycle 3 | 458.20 (103.355) | 1175.00 (117.331)
  Pre-dose on Day 1 Cycle 4: number analyzed (Participants) | 4 | 2
  Pre-dose on Day 1 Cycle 4 | 427.50 (83.636) | 678.50 (251.023)
  Pre-dose on Day 1 Cycle 5: number analyzed (Participants) | 0 | 1
  Pre-dose on Day 1 Cycle 5 |  | 819.00
  Pre-dose on Day 1 Cycle 7: number analyzed (Participants) | 1 | 2
  Pre-dose on Day 1 Cycle 7 | 243.00 | 621.50 (256.680)
  Pre-dose on Day 1 Cycle 10: number analyzed (Participants) | 1 | 1
  Pre-dose on Day 1 Cycle 10 | 334.00 | 759.00
  Pre-dose on Day 1 Cycle 11: number analyzed (Participants) | 0 | 1
  Pre-dose on Day 1 Cycle 11 |  | 770.00
  Pre-dose on Day 1 Cycle 13: number analyzed (Participants) | 1 | 1
  Pre-dose on Day 1 Cycle 13 | 267.00 | 807.00
  Pre-dose on EOT: number analyzed (Participants) | 1 | 1
  Pre-dose on EOT | 418.00 | 731.00
  Pre-dose on Safety Follow-up: number analyzed (Participants) | 4 | 4
  Pre-dose on Safety Follow-up | 101.93 (52.851) | 281.28 (241.454)

6. Secondary Outcome: Percentage of Participants With Transient Anti-Drug Antibody to Magrolimab - Safety Run-in (Part 1)
Time Frame: From Day 1 of Cycle 1 up to Safety Follow-up (30 days after last dose of magrolimab, maximum treatment duration 18.3 months); Cycle 1: 35 days, subsequent Cycles: 28 days.
Population: Immunogenicity Analysis Set included participants with at least one reported Anti-Drug Antibody result.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in)
Number analyzed (Participants) | 6 | 7
percentage of participants | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants With Objective Response According to Gynecologic Cancer InterGroup (GCIG) Criteria in Ovarian Cancer
Description: Objective response was defined as participants with a CR or a PR as assessed per GCIG criteria. The GCIG proposed use of both the RECIST and cancer antigen 125 (CA-125) criteria. A response according to CA-125 has occurred if there is ≥ 50% reduction in CA-125 levels from a pretreatment sample. The response had to be confirmed and maintained for at least 28 days. Participants can be evaluated according to CA-125 only if they had a pretreatment sample that was at least twice the upper limit of normal (ULN) and within 2 weeks prior to starting treatment. According to RECIST 1.1, CR was defined as disappearance of all target and all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (< 10 mm short axis). Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference baseline sum diameters.
Time Frame: as for outcome 3
Population: Participants in the Efficacy Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab 45 mg/kg + Avelumab 800 mg (Ovarian Cancer Participants)
Number analyzed (Participants) | 21
percentage of participants | 4.8 [0.1 to 23.8]

8. Secondary Outcome: Duration of Response (DOR) as Per GCIG Criteria in Participants With Ovarian Cancer
Description: DOR: time from initial response (CR or PR) until disease progression. Disease progression was defined according to RECIST 1.1 but can also be based on serum CA-125. Progression based on serum CA-125 levels was defined as (1) elevated CA-125 pretreatment and normalization of CA-125 with evidence of CA-125 ≥2x ULN on 2 occasions at least 1 week apart or; (2) elevated CA-125 pretreatment, which never normalizes, with evidence of CA-125 ≥2x nadir value on 2 occasions at least 1 week apart or; (3) CA-125 in normal range pretreatment with evidence of CA-125 ≥2x ULN on 2 occasions at least 1 week apart.
  Progression per RECIST 1.1: At least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum measured while on study (this included baseline sum if that was smallest). In addition to relative increase of 20%, sum must also demonstrate absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesion.
Time Frame: From initial response until disease progression or maximum time on study (26.2 months); assessed on Day 1 of Cycle 3 then every 2 cycles from Cycle 5 onwards up to 26.2 months; 1 cycle: 28 days
Population: Participants in the Efficacy Analysis Set who achieved objective response according to GCIG criteria. Only 1 participant was analyzed for this Outcome Measure. Data is not reported for participant confidentiality reasons.
Arm/Group | Magrolimab 45 mg/kg + Avelumab 800 mg (Ovarian Cancer Participants)
Number analyzed (Participants) | 0

9. Secondary Outcome: Progression-free Survival (PFS) in Participants With Ovarian Cancer
Description: PFS was defined as the duration of time from dose initiation to the first date of objectively documented disease progression per RECIST 1.1 or death, whichever occurred at first. Progression as per RECIST 1.1: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum measured while on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Participants who did not have documented disease progression and did not die were censored at their last tumor assessment date. Kaplan-Meier estimate was used for analysis
Time Frame: From first dose date to disease progression, death or maximum time on study (26.2 months); assessed on Day 1 of Cycle 3 then every 2 cycles from Cycle 5 onwards up to 26.2 months; 1 cycle: 28 days
Population: Participants in the Efficacy Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab 45 mg/kg + Avelumab 800 mg (Ovarian Cancer Participants)
Number analyzed (Participants) | 21
months | 2.0 [1.9 to 4.0]

10. Secondary Outcome: Overall Survival (OS) in Participants With Ovarian Cancer
Description: OS was defined as the duration of time from dose initiation to the date of death due to any cause. Participants who did not die were censored at their last known alive date.
  Kaplan-Meier estimate was used for analysis.
Time Frame: From first dose date to death or maximum time on study (26.2 months)
Population: Participants in the Efficacy Analysis Set were analyzed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab 45 mg/kg + Avelumab 800 mg (Ovarian Cancer Participants)
Number analyzed (Participants) | 21
months | 10.2 [2.1 to NA] — Upper limit of 95% confidence interval was not reached due to the low number of participants with events.

11. Secondary Outcome: Percent Change of Immune Cells by Immunohistochemistry in Participants With Ovarian Cancer
Description: Paired tumor biopsies from participants with ovarian cancer were analyzed by CD68 immunohistochemistry staining to evaluate the impact of magrolimab in combination with avelumab on macrophage frequency in the tumor microenvironment.
Time Frame: Screening and Day 1 Cycle 3 (Cycle 3 duration: 28 days)
Population: Participants who enrolled in ovarian cancer expansion cohort (Part 2) and for whom paired biopsies were available at both screening and Cycle 3 Day 1 were analyzed.
Measure: Mean (Full Range); unit: Percent Change
Groups:
- Magrolimab 45 mg/kg + Avelumab 800 mg (Part 2, Ovarian Cancer Expansion): Participants with checkpoint inhibitor-naïve ovarian cancer were treated with starting priming dose of 1 mg/kg of body weight magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1 followed by maintenance dose of 45 mg/kg of body weight magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15 and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles, in combination with 800 mg avelumab IV infusion (over 1 hour) on Days 8 and 22 of Cycle 1 and Days 1 and 15 of Cycle 2 and subsequent cycles.
Arm/Group | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 2, Ovarian Cancer Expansion)
Number analyzed (Participants) | 6
Percent Change | 137.8 [-66.67 to 700.0]

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose plus 30 days (maximum treatment duration 18.3 months) All-Cause Mortality: Enrollment up to 26.2 months
Description: Adverse Events: All treated participants included all participants who received at least 1 dose of any study drugs.
  All-Cause Mortality: All participants enrolled in study were analyzed. Per planned analysis, AE data were summarized by magrolimab maintenance dose level. One participant in Part 2 received maintenance dose of 20 mg/kg. Because of confidentiality reason, data for this participant was not provided separately and included in "Magrolimab Priming Dose or Magrolimab 20 mg/kg" arm.
Arm/Group | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in + Part 2, Ovarian Cancer Expansion) | Magrolimab Priming Dose or Magrolimab 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 5/6 | 10/25 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 15/25 | 2/3
Other Adverse Events (participants affected / at risk) | 6/6 | 25/25 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) (N=6) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in + Part 2, Ovarian Cancer Expansion) (N=25) | Magrolimab Priming Dose or Magrolimab 20 mg/kg (N=3)
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 4 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ammonia increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab 30 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in) (N=6) | Magrolimab 45 mg/kg + Avelumab 800 mg (Part 1, Safety Run-in + Part 2, Ovarian Cancer Expansion) (N=25) | Magrolimab Priming Dose or Magrolimab 20 mg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 8 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0
Photopsia (Eye disorders) | 1 | 2 | 0
Vitreous floaters (Eye disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 7 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 11 | 0
Vomiting (Gastrointestinal disorders) | 0 | 10 | 1
Asthenia (General disorders) | 0 | 3 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 3 | 9 | 1
Fatigue (General disorders) | 3 | 16 | 2
Influenza like illness (General disorders) | 0 | 3 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 14 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 11 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 6 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 7 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0
Headache (Nervous system disorders) | 4 | 16 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-12-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT03558139/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT03558139/SAP_001.pdf